CLINICAL TRIAL: NCT04405284
Title: Disinfection Practices Among Women in Egypt During the Coronavirus Pandemic.
Brief Title: The Use of Disinfectants Among Women in Egypt and the Toxicity by Bleach During the Coronavirus Lock-down.
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Maha Farid,MBBCh, MSc,PhD, Lecturer in the department of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Helwan University
Other Study IDs: COVID2020_HelwanU_01
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Toxicity by Bleach
Keywords: women; Egypt; disinfectatnts; adverse reactions; coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: use and exposure to disinfectants during the coronavirus pandemic — The use of disinfecting products in deep house cleaning by women during the coronavirus lockdown.

SUMMARY:
This study examines the use of disinfectants by Egyptian women during the coronavirus lockdown. Data will be collected via an online self-administered questionnaire that will be distributed to Egyptian women via social media channels. Questions in the questionnaire will assess types of disinfectants frequently used and how often they have been used for household disinfection during the 2020 coronavirus pandemic. The investigators hypothesized that the frequent use of disinfectants in deep household cleaning during the lockdown has been associated with increased incidents of toxicity by bleach and similar products. At the same time, people were advised to stay home and refrain from seeking in-person medical care to avoid catching the coronavirus. Therefore, many people used social media to receive medical advice not necessarily from the right sources nor qualified experts.

DETAILED DESCRIPTION:
This study examines the use of disinfectants by Egyptian women during the coronavirus lockdown. Data will be collected via an online self-administered questionnaire that will be distributed to Egyptian women via social media channels such as (Facebook and WhatsApp).

Google Forms tool will be used to conduct the questionnaire as questions in the questionnaire will assess types of disinfectants frequently used and how often they have been used for household disinfection during the 2020 coronavirus pandemic. Questions will also assess the occurrence of adverse effects related to the increased use of disinfectants during the lockdown and how women reached out for medical care for their family members in cases of accidental toxicity.

The investigators hypothesized that the frequent use of disinfectants in deep household cleaning during the lockdown has been associated with increased incidents of toxicity by bleach and similar products. At the same time, people were advised to stay home and refrain from seeking in-person medical care to avoid catching the coronavirus. Therefore, many people used social media to receive medical advice not necessarily from the right sources nor qualified experts.

The questionnaire is designed by the primary investigator (Dr. Maha Farid) and was reviewed by other experts in the field of forensic medicine and clinical toxicology. The questions were developed in English and then translated in Arabic to be distributed to the target population in Arabic.

The inclusion criteria for women participating in this survey will include adult females living in Egypt during the time of lockdown due to coronavirus pandemic that started in Egypt in March 2020.

The questionnaire will be open for a month or till we reach the desired sample size, whichever comes first.

The data collected via this questionnaire will be then tabulated and analyzed using the proper statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult women living in Egypt the coronavirus lockdown started in March 2020

Exclusion Criteria

* Men living in Egypt
* Adult women not living in Egypt during the coronavirus lockdown started in March 2020.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aging 18 years old and above located in Egypt during the coronavirus lockdown in March 2020.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
The use of disinfectants in deep house cleaning by women in Egypt. | one month after the distribution of the questionnaire
  Assessment of disinfection practice among women in Egypt

CONTACTS AND LOCATIONS:
Overall Officials: Maha M Farid, PhD, Principal Investigator — Helwan University
Locations (1):
- Maha M Farid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The plan to make (IPD) viable has not been decided to maintain the confidentiality and privacy of the information collected in this research project.